CLINICAL TRIAL: NCT02557581
Title: cAMP Signaling and Muscle Adaptations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Nielsen, Post.Doc, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: TUD
Record Dates: First submitted 2015-09-13; First posted 2015-09-23 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Muscle Hypertrophy in Healthy Young Men
MeSH Terms: interventions — Endurance Training; Resistance Training; Terbutaline; Clenbuterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Terbutaline (Experimental): Beta2-adrenergic stimulation with terbutaline
  Interventions: Other: No training; Other: Endurance training; Other: Resistance Training; Drug: Terbutaline
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: No training; Other: Endurance training; Other: Resistance Training; Drug: Placebo
- Clenbuterol (Experimental): Beta2-adrenergic stimulation with clenbuterol
  Interventions: Other: No training; Drug: Clenbuterol

INTERVENTIONS:
Other: No training
Other: Endurance training
  Arms: Placebo; Terbutaline
Other: Resistance Training
  Arms: Placebo; Terbutaline
Drug: Terbutaline
  Arms: Terbutaline
Drug: Clenbuterol
  Arms: Clenbuterol
Drug: Placebo
  Arms: Placebo

SUMMARY:
The role of cAMP signaling mediated by beta2-adrenergic stimulation with agonists has been well-studied in skeletal muscles of animals. Studies in humans are scant and the scope of the present study is thus to investigate the role of cAMP signaling by beta2-adrenergic stimulation for muscle adaptations in humans.

ELIGIBILITY:
Inclusion Criteria:

* healthy young men
* 18-35 years of age
* Informed consent
* Active 2-5 hours of training pr. week
* Maximal oxygen uptake (ml/min/kg) of 40-60
* Lean body mass of 55-65 kg / Lean mass index 14-22 kg/m2

Exclusion Criteria:

* Smoker
* Allergy towards study drugs
* Chronic disease

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-06-30 (Actual); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Muscle hypertrophy (lean body mass in Kilograms) | 2 days
  Lean body mass (kg) will be measured at two different days by Dual X-ray absorbance (DXA)

SECONDARY OUTCOMES:
Energy turnover (ml/min or mmol/kg dry weight muscle) | 1 day
  Pulmonary gas exchange and lactate and glycogen will be measured in muscle biopsies obtained before and after intense exercise

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of Nutrition, Exercise and Sports, Copenhagen
  - Bispebjerg University Hospital, Copenhagen